CLINICAL TRIAL: NCT00732030
Title: Evaluation of the Acrysof Toric Model SN60T3 Intraocular Lens in Patients With Predicted Residual Corneal Astigmatism Between 0.75 and 1.03 Diopters (D)
Brief Title: Low Cylinder Toric
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin/Director - Global Scientific Market Affairs, Alcon Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M07-005
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2010-04-07 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-03

CONDITIONS: Cataracts
Keywords: Toric IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AcrySof Toric T3 (Experimental): Each enrolled eye receives AcrySof Toric Model SN60T3 Intraocular Lens (IOL)
  Interventions: Device: Toric IOL (SN60T3)

INTERVENTIONS:
Device: Toric IOL (SN60T3) — Each enrolled eye implanted with the AcrySof Toric Model SN60T3 intraocular lens (IOL) for the treatment of cataract.

SUMMARY:
Study evaluates the visual outcomes and patient satisfaction after implantation of a toric intraocular lens (IOL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cataracts
* Predicted residual corneal astigmatism between 0.75 and 1.03 Diopters (D)

Exclusion Criteria:

* Preoperative ocular pathology
* Planned monovision

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were >21 years of age, of any race and either gender. Patients had operable cataracts in at least 1 eye and were able to provide informed consent. Patients were free of systemic diseases affecting ocular health and had a predicted residual corneal astigmatism between 0.75 and 1.03 Diopters (D) by the AcrySof Toric calculator.
Pre-assignment Details: During the preoperative exam, subjects were examined to ensure they met the inclusion/exclusion criteria. Only subjects who signed an informed consent and qualified to be in the study by meeting all inclusion/exclusion criteria were enrolled.
Groups:
- AcrySof Toric T3: Each enrolled eye receives AcrySof Toric SN60T3 IOL
Period: Overall Study
Arm/Group | AcrySof Toric T3
Started | 26
Completed | 24
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | AcrySof Toric T3
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Distance Visual Acuity
Description: Uncorrected Distance Visual Acuity at month 6 measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". It is a unit of measure for visual acuity (VA).
Time Frame: 6 months
Population: Data was collected for 29 eyes in 24 patients.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | AcrySof Toric T3
Number analyzed (Participants) | 24
logMAR | 0.09 (0.14)

2. Primary Outcome: Best Corrected Distance Visual Acuity
Description: Best Corrected Distance Visual Acuity at month 6 measured in LogMAR. LogMAR is the "logarithm of the minimum angle of resolution". It is a unit of measure for visual acuity (VA).
Time Frame: 6 Months
Population: Data was collected for 29 eyes in 24 patients.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | AcrySof Toric T3
Number analyzed (Participants) | 24
logMAR | 0.02 (0.09)

3. Primary Outcome: Residual Refractive Cylinder
Description: Residual Refractive Cylinder at month 6 measured in diopters (D).
Time Frame: 6 Month
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | AcrySof Toric T3
Number analyzed (Participants) | 24
Diopters | 0.4 (0.4)

4. Secondary Outcome: Patient Satisfaction Survey
Description: Satisfaction for daytime distance vision, nighttime distance vision, and indoors distance vision on a scale of 1 to 5, with 1 being very dissatisfied and 5 being very satisfied.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | AcrySof Toric T3
Number analyzed (Participants) | 24
Units on a Scale
  Daytime Distance Vision | 4.6 (0.6)
  Nighttime Distance Vision | 4.4 (0.7)
  Indoors Distance Vision | 4.6 (0.7)

ADVERSE EVENTS:
Time Frame: Surgical visit through 6 month postoperative visit.
Arm/Group | AcrySof Toric T3
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written agreement.